CLINICAL TRIAL: NCT02230605
Title: Perioperative Cognitive Protection - Cognitive Exercise and Cognitive Reserve (The Neurobics Trial)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Michelle Humeidan, Assistant Professor of Clinical Anesthesiology, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2013H0388
Record Dates: First submitted 2014-08-29; First posted 2014-09-03 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Delirium
Keywords: Delirium; Post Operative Delirium; PD; POD; Anesthesia; Anesthesiology; Post Operative Recovery; Post Anesthesia Care Unit; PACU; Cognition; Cognitive Impairment; Memory; Thinking; Confusion Assessment Method; CAM; Neurobics; Neuroplasticity; Lumosity; Brain Games; Cognitive Exercise; Cognitive Training; Perioperative Cognitive Protection; Cognitive Reserve; Neurobics Trial; Surgery; Elderly Patients
MeSH Terms: conditions — Delirium; Emergence Delirium; Cognitive Dysfunction | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Exercise (Experimental): The cognitive exercises will consist of a series of computer games focusing on five categories: memory, speed, attention, flexibility and problem-solving. Participants will be expected to complete 1 hour of Lumosity exercise daily for a minimum of 8 days prior to surgery. Participants will be instructed to complete no less than 15 minutes of exercise at a time throughout each day. Each hour of exercise, participants will work through at least 1 game under each category. Research assessments will include Mini-Mental State Examination, Self-Administered Gerocognitive Examination, Geriatric Depression Scale, Charlson Comorbidity Index, Short Form 36 Health Survey, Confusion Assessment Method, Memorial Delirium Assessment Scale and Postoperative Quality of Recovery Scale.
  Interventions: Other: Mini-Mental State Examination; Other: Self-Administered Gerocognitive Examination; Other: Geriatric Depression Scale; Other: Charlson Comorbidity Index; Other: Short Form 36 Health Survey; Other: Confusion Assessment Method; Other: Memorial Delirium Assessment Scale; Other: Postoperative Quality of Recovery Scale
- Normal Activity (Placebo Comparator): Participants randomized into the Normal Activity group will be encouraged to maintain their normal activity level prior to surgery. These participants are asked not to alter their normal daily routine of mental exertion (i.e. watching television, reading, puzzles, etc.) and not permitted to subscribe to Lumosity while in the research study. Research assessments will include Mini-Mental State Examination, Self-Administered Gerocognitive Examination, Geriatric Depression Scale, Charlson Comorbidity Index, Short Form 36 Health Survey, Confusion Assessment Method, Memorial Delirium Assessment Scale and Postoperative Quality of Recovery Scale.
  Interventions: Other: Mini-Mental State Examination; Other: Self-Administered Gerocognitive Examination; Other: Geriatric Depression Scale; Other: Charlson Comorbidity Index; Other: Short Form 36 Health Survey; Other: Confusion Assessment Method; Other: Memorial Delirium Assessment Scale; Other: Postoperative Quality of Recovery Scale

INTERVENTIONS:
Other: Mini-Mental State Examination — To be completed at the Screening Visit and Post-Operative Day 7 Visit (or Discharge)
  Other Names: MMSE
Other: Self-Administered Gerocognitive Examination — To be completed at the Screening Visit and Post-Operative Day 7 Visit (or Discharge)
  Other Names: SAGE
Other: Geriatric Depression Scale — To be completed at the Screening Visit and at POD 90
  Other Names: GDS
Other: Charlson Comorbidity Index — To be completed at the Screening Visit and at POD 90
  Other Names: CCI
Other: Short Form 36 Health Survey — To be completed at the Screening Visit
  Other Names: SF-36
Other: Confusion Assessment Method — To be completed at the Day 0 (Pre-Operative) Visit, Day 0 (Post-Operative) Visit, and Day 1-7 Visits at 7:30AM ± 1.5 hrs and 6:30PM ± 1.5 hrs. (or until hospital discharge)
  Other Names: CAM
Other: Memorial Delirium Assessment Scale — To be completed at the Day 0 (Pre-Operative) Visit, Day 0 (Post-Operative) Visit, and Day 1-7 Visits at 7:30AM ± 1.5 hrs and 6:30PM ± 1.5 hrs. (or until hospital discharge)
  Other Names: MDAS
Other: Postoperative Quality of Recovery Scale — To be completed at Day 0 (Post-Operative) Visit, and Day 1-7 Visits at 6:30PM ± 1.5 hrs (or until hospital discharge). Will be completed POD 7 over the phone if patient already discharged. Will be completed on POD 30 and POD 90.
  Other Names: PQRS

SUMMARY:
Many individuals experience an acute change in thinking and reasoning skills after surgery. This is called post-operative delirium (PD). PD symptoms typically start 1-3 days after surgery. Advanced age has been identified as a risk factor for PD. The purpose of this study is to determine if performing mental exercise, before surgery, will help reduce post-surgery memory and thinking problems. Assuming a 30% incidence of PD and proposed 50% reduction of PD in the intervention group (15% incidence), a total of 242 patients (1:1 ratio, 121 in each group) will achieve 80% power to detect 50% reduction using chi-square test at a 5% type I error rate. Assuming approximately 1/3 of consented patients either fail screening or do not complete the study after consent, we expect to consent 358 patients.

At least 8 days before surgery, subjects complete a series of questionnaires to assess baseline cognition level (or thinking ability) and status of overall well-being. At the completion of the screening visit, qualifying subjects are randomized into two groups:

Participants randomized into the Cognitive Exercise group are expected to complete tablet-based brain games provided by Lumosity. These subjects are given a handheld tablet for the duration of the preoperative period. Participants in this group are expected to complete a minimum of 10 hours within at least 8 days prior to surgery.

Participants randomized into the Normal Activity group are encouraged to carry out their baseline daily activities, and do not have any study-related cognitive exercise expectations before surgery. These subjects still complete the same questionnaires and assessments as the Cognitive Exercise group throughout the study, however, are asked not to alter their normal daily routine of mental exertion (i.e. watching television, reading, puzzles, etc.) and are not permitted to subscribe to Lumosity while in the research study.

On the day of surgery, a baseline delirium evaluation (CAM - Confusion Assessment Method) is taken before surgery. During surgery, research personnel monitor vital signs and medications given. After surgery, another CAM evaluation is taken in the post-operative recovery room.

Throughout the subject's hospital stay, pain levels and medication usage are recorded. The CAM and MDAS (Memorial Delirium Assessment Scale) are used to identify and determine severity of PD. The evaluations are given twice daily, at at 7:30AM ± 1.5 hrs and 6:30PM ± 1.5 hrs, for 7 days or until hospital discharge (whichever comes first). The Postoperative Quality of Recovery Scale (PQRS) is used each post-operative day at 6:30PM ± 1.5 hrs until discharge, and completed over the phone on POD 7 if patient discharged. The PQRS is also administered over the phone on POD 30 and POD 90.

DETAILED DESCRIPTION:
Potential study participants will be identified one of two ways, either by the treating physician in clinic when the decision is made to pursue surgery or by researchers monitoring the OR schedule. When a potential participant is identified by the treating physician in clinic, they will ask the patient if study personnel may call them to discuss the study. If the patient agrees to be contacted, the surgeon will alert study personnel who will call the patient to explain the study and arrange the initial study (screening) visit. Study personnel will monitor the OR schedule and call any potential patients the surgeons have not already identified in clinic. In this case, patients will be informed over the phone that their surgeon has granted permission to contact them regarding the study. Surgeons will be made aware when their patients have been approached over the phone, and updated accordingly if the patient agrees to the screening visit and is subsequently enrolled in the study. All screening visits will occur at the OSU Pre-operative Assessment Center (OPAC). When possible the screening visit will co-inside with pre-operative testing per the Anesthesia Department at OPAC.

Informed consent will occur at the initial screening visit which is to take place approximately 2 weeks prior to surgery, but no less than 8 days pre-op. At this visit, a member of the research team will obtain demographic information (gender, education level), historical medical information, and information regarding medication usage. The researcher will perform the Mini-Mental Status Exam (MMSE) - the modified version (see attached document), Self Administered Gerocognitve Form (SAGE) - all four versions (see attached questionnaires), Geriatric Depression Scale, Charlson Comorbidity Index, Postoperative Quality Recovery Scale (PQRS), and Short-form 36 Health Related Quality of Life Measure. Patients meeting inclusion criteria will be randomized to either the cognitive exercise or control group. Patients in the cognitive exercise group will be given a tablet with preinstalled access to Lumosity (Lumos Labs, San Francisco, CA, USA), a cognitive exercise software application which will be used in this study. Each participant in the cognitive exercise group will be expected to complete 1 hour of Lumosity brain exercise daily for a minimum of 8 days prior to surgery, equaling an effective 'dose' at least 10 hours. Playing time will be determined either by: (a) the actual in-game playing time; or (b) as calculated by the research team during the Screening Visit (see the "Subject Diary"). The Lumosity software allows for monitoring of participant compliance by researchers. Patients in the control group will carry out their normal activities prior to surgery.

All patients will undergo surgery as planned. On the day of surgery, prior to proceeding to the operating room, patients will be assessed with the Confusion Assessment Method (CAM) to confirm no presence of delirium pre-operatively. In the Post-anesthesia Recovery Unit, a different member of the research team (blinded to the patient's group assignment) will repeat the CAM to assess for PD. While hospitalized, pain scores determined using the Verbal Analog Scale and narcotic use will be obtained from the electronic medical record with at least 8 hour frequency (entered by registered nurses). All participants will be evaluated by a blinded researcher using the combined CAM/Memorial Delirium Assessment Scale (MDAS) at 7:30AM ± 1.5 hrs and 6:30PM ± 1.5 hrs for PD on subsequent post-op days until discharge. Additionally, the PQRS will be completed at each 6:30PM ± 1.5 hrs assessment. The PQRS, MMSE, and SAGE will be repeated just prior to discharge or on POD 7. A different form for the SAGE examination, as well as alternate number and word sequences for the PQRS and MMSE assessments, will be used in order to reduce the potential influence of the learning effect. At the end of this visit, active patient participation is complete. For subjects discharged before POD 7, the PQRS will be given again via telephone. Follow-up visits will be conducted on POD 30 and POD 90 via telephone. The PQRS will be obtained on POD 30, and the PQRS, GDS, and SF-36 will be obtained on POD 90. The research team will also periodically check the medical record during this time for readmissions and provider notes related to medical events. Participation is complete after POD 90.

ELIGIBILITY:
Inclusion Criteria

1. 60 years of age or older
2. Capable and willing to consent
3. Non-cardiac/non-neurological surgery with expected hospital stay of at least 72 H
4. American Society of Anesthesiologists (ASA) physical status I-IV
5. English speaking
6. Willingness to use a provided tablet device
7. Willingness to commit at least 1 hour per day to experimental intervention (cognitive activity/exercise) to complete a minimum of 10 hours within at least 8 days prior to surgery.

Exclusion criteria

1. Severe visual or auditory deficits
2. Illiterate
3. Surgery within the previous 6 months requiring general anesthesia
4. Score < 26 on initial Mini Mental Status Exam (MMSE - modified version) (24 for patients with less than high school education)
5. Positive pre-surgery Confusion Assessment Method test (CAM)
6. Active depression as indicated by Geriatric Depression Scale screening test (score ≥ 10)
7. History of Axis I or II psychiatric disorders including bipolar disorder, schizophrenia, dementia, alcohol or drug abuse
8. ASA physical status V, VI
9. Planned postoperative intubation

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2015-07; Primary Completion 2019-05-20 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
Reduction in the incidence of Post-Operative Delirium (%) | Post-Operative Period (Day 0 through Day 7 or Discharge, whichever comes first)
  Assuming a 30% incidence of PD and proposed 50% reduction of PD in the intervention group (15% incidence), a total of 242 patients (1:1 ratio, 121 in each group) will achieve 80% power to detect 50% reduction using chi-square test at a 5% type I error rate. Assuming approximately 1/3 of consented patients either fail screening or do not complete the study after consent, we expect to consent 358 patients. The incidence of PD will be compared between the control group and the intervention group as detected by the Confusion Assessment Method (CAM) / Memorial Delirium Assessment Scale (MDAS). Once a patient is positive, they will no longer be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle L Humeidan, MD,PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Humeidan ML, Reyes JC, Mavarez-Martinez A, Roeth C, Nguyen CM, Sheridan E, Zuleta-Alarcon A, Otey A, Abdel-Rasoul M, Bergese SD. Effect of Cognitive Prehabilitation on the Incidence of Postoperative Delirium Among Older Adults Undergoing Major Noncardiac Surgery: The Neurobics Randomized Clinical Trial. JAMA Surg. 2021 Feb 1;156(2):148-156. doi: 10.1001/jamasurg.2020.4371. PMID 33175114
- [Derived] Humeidan ML, Otey A, Zuleta-Alarcon A, Mavarez-Martinez A, Stoicea N, Bergese S. Perioperative Cognitive Protection-Cognitive Exercise and Cognitive Reserve (The Neurobics Trial): A Single-blind Randomized Trial. Clin Ther. 2015 Dec 1;37(12):2641-50. doi: 10.1016/j.clinthera.2015.10.013. Epub 2015 Nov 17. PMID 26598177